CLINICAL TRIAL: NCT04915820
Title: Iron and Vaccine-preventable Viral Disease
Brief Title: Iron and COVID-19 Vaccine Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Prof Simon Karanja, PhD, Jomo Kenyatta University of Agriculture and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DIVA I
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2021-09

CONDITIONS: Iron Deficiency Anemia; Vaccine Response Impaired; COVID-19 Vaccine; Iron Deficiency Anemia Treatment
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate iron treatment (Active Comparator): intravenous iron carboxymaltose before vaccination
  Interventions: Dietary Supplement: Ferinject
- No iron treatment (No Intervention): no intravenous iron carboxymaltose before vaccination

INTERVENTIONS:
Dietary Supplement: Ferinject — intravenous iron carboxymaltose
  Arms: Immediate iron treatment

SUMMARY:
Vaccines often underperform in Africa compared to high-income countries. Why vaccines do not work as well in Africa remains uncertain. Malnutrition likely plays a role. Our study objective is to assess whether iron deficiency anaemia in young women impairs their immune response to the COVID-19 vaccine, and whether iron treatment improves their response.

DETAILED DESCRIPTION:
Group 1 (immediate iron treatment) will receive iron treatment before vaccination. Women in both groups will receive the 1st dose of the COVID-19 vaccine. Vaccine response will be measured 28 and 56 days after the first vaccine administration in both groups. At 28 days, participants will receive the 2nd dose of the COVID-19 vaccine. Group 2 (delayed iron treatment) will receive iron treatment at study end.

ELIGIBILITY:
Inclusion Criteria:

18-55 years old Zinc protoporphyrin > or equal 40 mmol/mol heme hemoglobin < or equal 109 g/L no malaria no known HIV infection no medical condition that precludes study involvement no iron supplementation 1 week prior to study start no recent tuberculosis infection no vaccination of yellow fever or influenza prior to enrolment not pregnant

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Antibody titers | day 35
Antibody titers | day 63
Seroconversion | day 35
Seroconversion | day 63
Antibody avidity index | day 35
  percentage of antibodies that remain bound to beads
Antibody avidity index | day 63
  percentage of antibodies that remain bound to beads

SECONDARY OUTCOMES:
antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response | day 0
  immunoassay
antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response | day 7
  immunoassay
antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response | day 35
  immunoassay
antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response antiviral immunoglobulin G response | day 63
  immunoassay
immune cell populations | day 0
  number and type of immune cells
immune cell populations | day 7
  number and type of immune cells
immune cell populations | day 35
  number and type of immune cells
immune cell populations | day63
  number and type of immune cells
Proteomics | day 0
  Proteins involved in immune response
Proteomics | day 7
  Proteins involved in immune response
Proteomics | day 35
  Proteins involved in immune response
Proteomics | day 63
  Proteins involved in immune response
Transcriptomics | day 0
  Genes involved in immune response
Transcriptomics | day 7
  Genes involved in immune response
Transcriptomics | day 35
  Genes involved in immune response
Transcriptomics | day 63
  Genes involved in immune response
Immune cell cytokine secretion | day 7
  ELISpot
Immune cell cytokine secretion | day 35
  ELISpot
Hemoglobin | day 0
  iron status parameter
Hemoglobin | day 7
  iron status parameter
Hemoglobin | day 35
  iron status parameter
Hemoglobin | day 63
  iron status parameter
Plasma ferritin | day 0
  iron status parameter
Plasma ferritin | day 7
  iron status parameter
Plasma ferritin | day 35
  iron status parameter
Plasma ferritin | day 63
  iron status parameter
Transferrin receptor | day 0
  iron status parameter
Transferrin receptor | day 7
  iron status parameter
Transferrin receptor | day 35
  iron status parameter
Transferrin receptor | day 63
  iron status parameter
Transferrin saturation | day 0
  iron status parameter
Transferrin saturation | day 7
  iron status parameter
Transferrin saturation | day 35
  iron status parameter
Transferrin saturation | day 63
  iron status parameter
C-reactive protein | day 0
  inflammation status parameter
C-reactive protein | day 7
  inflammation status parameter
C-reactive protein | day 35
  inflammation status parameter
C-reactive protein | day 63
  inflammation status parameter
Alpha-glycoprotein | day 0
  inflammation status parameter
Alpha-glycoprotein | day 7
  inflammation status parameter
Alpha-glycoprotein | day 35
  inflammation status parameter
Alpha-glycoprotein | day 63
  inflammation status parameter
retinol binding protein | day 0
  vitamin A status marker
retinol binding protein | day 7
  vitamin A status marker
retinol binding protein | day 35
  vitamin A status marker
retinol binding protein | day 63
  vitamin A status marker
plasma zinc | day 35

CONTACTS AND LOCATIONS:
Overall Officials: Simon Karanja, PhD, Principal Investigator — JKUAT Nairobi
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya